CLINICAL TRIAL: NCT04613583
Title: Normal Development of the Human Fetus and the Influences and Mechanisms by Which That Development Occurs and is Perturbed
Brief Title: Scottish Advanced Fetal Research Study
Acronym: SAFeR
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Principal Investigator, Paul A Fowler, Director of the Institute of Medical Sciences, University of Aberdeen
Other Study IDs: 2-051-15
Record Dates: First submitted 2017-12-19; First posted 2020-11-03 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Fetal Developmental Abnormality; Fetal Development; Human; Life Style
Keywords: fetal; human; gestation; development; congenital; exposures; maternal; life style; exogenous chemicals; obesity; deprivation; alcohol; cigarette; endocrine disruption
MeSH Terms: conditions — Congenital Abnormalities; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Human fetal blood and multiple organs (including brain, heart, lungs, liver, skin, joints, gonads, urogenital system, pancreas, thyroids, adrenals)
  Placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SAFeR Fetuses: Different maternal lifestyle factors: smoking, BMI, social deprivation, alcohol use, medicines. Depends on specific subproject analyses.
  Interventions: Other: SAFeR fetuses

INTERVENTIONS:
Other: SAFeR fetuses — NO active intervention performed.

SUMMARY:
In-utero exposure to drugs and chemicals through maternal smoking, alcohol use, drug abuse, prescription medicines and occupational/lifestyle exposures is widespread. Such exposures can alter fetal development and programming, leading to the effects becoming "locked in" from birth and causing long-term adverse consequences for the individual. These include costly and widespread conditions such as obesity, hypertension, metabolic syndrome and infertility. The weight of evidence linking these conditions to fetal recreational drug or environmental chemical exposures, including cigarettes, alcohol, air pollution, food contact materials, is overwhelming. What is lacking is an understanding of how fetal drug exposure translates to adult ill-health and this is due, largely, to an inability to study the problem directly in affected human fetuses. The investigators, and others, have shown that human fetal development, which lays the foundations of adult health and function (fetal programming), is quite different from the rodent and frequently exhibits surprising aspects. It has become evident that the close interconnectivity of the developing fetal organs and also the placenta, means that a much more holistic approach to research aiming to understand human fetal development and the challenges posed to programming for a health adulthood is critical. To that end the investigators have established a carefully considered gestational age range (7-20 weeks of gestation) of fetuses we can study together with multiple fetal organs and body fluids collected and maternal information recorded.

The overarching objective of the study is to intensively and systematically study the human fetus during a normal pregnancy and pregnancies where aspects of maternal lifestyle and environment will challenge the fetus. The investigators aim to provide fundamental information to better understand the mechanisms involved and to detect and treat or ameliorate adverse effects during pregnancy (such as maternal smoking/drinking, deprivation, exposure to pollution). In the long term findings from this research will be important for future studies aimed at enabling better health in later life.

DETAILED DESCRIPTION:
Primary Objective

To provide fundamental information to better understand the mechanisms involved and to detect and treat or ameliorate adverse effects during pregnancy.

Secondary Objectives

The secondary objectives of this study are aimed at better understanding of normal processes during development and how maternal lifestyle and environment can affect it. The investigators' research will involve a wide range of laboratory, cell and tissue culture and xenografting as well as microscopic techniques to study chemicals, hormones, proteins, genes and DNA in the fetal tissues. The investigators have developed sophisticated approaches to minimise how much tissue is required to carry out as many different measurements as possible in the same sample. It should be noted that the proposed studies are collaborative with different research groups since no single research group could carry out all the studies in isolation. Furthermore, the proposed studies will inform back to animal and cell studies, enabling more accurate interpretation of their own findings in light of mechanisms and specific conditions actually at play in the human fetus.

1. Human fetal endocrine system

   The investigators aim to investigate how the different hormone systems in the fetus develop and are affected by adverse maternal factors such as cigarette smoking and obesity. These include the testis, ovary, adrenal gland, thyroid gland, kidney and the hypothalamus, pineal gland and pituitary gland in the brain. In addition, the investigators also aim to study the placenta, including its endocrine function, and how it is affected by maternal environment, since it is a key organ of pregnancy. Changes in programming that establishes the endocrine system can have lifelong consequences for health and wellbeing.
2. Human fetal reproductive and urogenital system

   The investigators aim to investigate how the ovary, testis, urogenital tract (including prostate gland, breast buds and uterus), genitalia and kidney develop in the human fetus. There is considerable evidence that maternal smoking and over the counter medicine use can have negative impacts on this system and we will investigate when such impacts begin and what mechanisms are involved. In addition, common cancers, such as testis cancer, may have fetal origins and certainly events in fetal life may predispose the resulting adult to develop cancers. In the case of testis, ovary, breast buds and prostate gland, an additional aim is to determine whether and how events between 7 and 20 weeks of gestation increase the likelihood of cancers in these organs in adulthood.
3. Mechanistic studies, Epilepsy and other brain disorders

   The investigators aim to investigate development of the fetal central nervous system, including the brain. The first study planned is to investigate changes in genes and the structure of DNA in the brain related to epilepsy and other neurodevelopmental disorders linked with maternal cigarette smoking during pregnancy. A second aim is to use the smoke-exposed fetuses to better understand the role vitamin A plays in normal fetal development, including development of the central nervous system. Similar concerns are expressed in the literature with respect to maternal alcohol consumption and by accessing data from the Fast Alcohol Screening Test alcohol questionnaire that is already collected at clinic, the investigators will be able to address this issue systematically with respect to all the studies, including fetal brain development.
4. Metabolism and liver disease

   The investigators aim to continue their studies (funded by the Medical Research Council) of the human fetal liver and other organs important for metabolism, including pancreas and fat cells and cells that will become fat cells (precursor cells). Programming of metabolism during life in the womb is important for adult health and better understanding of the development of the metabolic systems and how they are perturbed by factors such as maternal smoking and deprivation is an important basis of developing strategies for wellbeing post-natally. A critical disease of growing importance in these studies is non-alcoholic fatty liver disease, which is increasing in incidence, especially in obese individuals. Given that the human fetal liver is active and responding to maternal environment, some of the basis of this disease may be established in fetal life. In addition, the development of thyroid and adrenal glands is also essential in establishing normal metabolic processes. Cutting edge techniques, such as large-scale metabolomic and lipidomic studies, including analysis of a wide range of dietary metabolites, will also be used.
5. Heart and cardiovascular system

   The development of the heart and the major artery, the aorta, between 7 and 20 weeks of gestation will be characterised. The effects of adverse in-utero environment of the developmental processes will then be investigated.
6. Immune system development

   The thymus is critical and large organ in fetal development that is important to establish the immune system. The spleen manufactures antibodies and, in fetal life, red blood cells (as does the fetal liver) and recycles red blood cells. Both organs have important role in maintaining the immune system. The investigators aim to investigate whether adverse maternal lifestyle and/or environment can alter thymus and spleen development and function.
7. Bone, cartilage and joints

   Very little is known about normal bone and cartilage development in the human fetus. Importantly, it is not even know when the cells involved in bone, cartilage and joint development begin to alter their behaviour into a more "adult" format. The reason this is important is that in musculoskeletal disease in the elderly, especially osteoarthritis, early stages of disease is usually characterised by renewed tissue growth - i.e. a return to a more "fetal" pattern of cell behaviour. The role of cell programming during fetal life and better understanding of the correct development and maintenance of bone, cartilage and joints, and how programming is affected by the fetal environment, is therefore one of the investigators' aims.
8. The development of the placenta between 7 and 20 weeks of gestation

   A great deal is known about the term placenta because it is so easy to obtain and to relate directly to the accompanying new-born and its parents. However, the placenta is a dynamically developing organ that is vital for normal pregnancy and that is affected by maternal lifestyle (e.g. placental growth is reduced if the mother continues to smoke while pregnant). The investigators aim therefore to better understand how the placenta develops during this window in gestation and how it is affected by maternal environment.
9. Nerve repair

   Spinal cord injury is a massive health problem globally. Recently it has been shown that human fetal central nervous system cells or embryonic nerve stem cells have the potential to assist in novel treatment strategies to repair spinal cord injury. This final secondary objective is focussed on a proof of concept study to determine whether culturing severed nerves in the presence of human fetal nerve cells assists in correct and functional nerve regrowth and re-joining across the induced gap. Any further studies, if the proof of concept aim is realised in a satisfactory manner would require a separate ethic application.
10. Maternal emotional health and wellbeing effects on the fetus

    Maternal stress is a well-known negative influence on fetal development. The investigators' aim is to perform a pilot study relating indices of fetal development, such as morphology, endocrine status, to maternal records of emotional health and wellbeing and abuse. The principal outcome will be an indication as to whether maternal stress is affecting fetal development at a general level between 7 and 20 weeks of gestation. Placental biomarkers identified in other studies listed above will also be related to measures of maternal stress in order to establish whether there may be placental biomarkers of early fetal response to maternal stress.
11. Fetal lung

    While it is well known that the adverse effects of maternal smoking include increased incidences of respiratory problems, such as asthma. However, there are also data suggesting that the offspring exposed to cigarette smoke may be more likely to develop lung cancer. The investigators' aim is to determine whether maternal smoking disturbs fetal lung development early in pregnancy and if this includes signs of increased likelihood of cancer development, such as polycyclic aromatic hydrocarbon-DNA adducts in the fetal lungs.
12. Quantifying human fetal exposure to pollutants, drugs, pharmaceuticals and other chemicals

    It is simple to measure chemicals in the blood or urine of the mother, or in amniotic fluid collected during amniocentesis. However, amniocentesis is not performed for research purposes because of not inconsiderable risk to the fetus. This means reliance on animal studies of such chemicals getting to the fetus but this is rather inadequate due to major species differences. Therefore the investigators aim to measure chemicals and drugs of potential health concern (such as bisphenol A which is in plastics and over the counter drugs taken by mothers which may affect the fetus, such as paracetamol) in the fetal tissues, including blood and urine where available. This is the only way to accurately assess how much of these compounds actually get into the fetus itself. This is important since the fetus is considered much more vulnerable than the adult to toxic chemicals. In addition, the investigators aim to also measure these compounds in the placentas (and cord blood where available) from the same fetuses. Because the placenta is readily available at term, placental biomarkers of fetal exposure to adverse compounds (e.g. alcohol) that are detected in the second trimester fetal liver will be investigated in the term placenta.
13. Non-genetic programming of the fetus for adult life

Epigenetic changes are changes that involve marks being put onto DNA that affects how genes are activated. Therefore, an epigenetic change can change, sometimes greatly, the link between the amount of a gene present in cell and its effect. This linkage can be quite large with a gene being practically silenced in terms of its effect, even though there may be plenty of the gene present in the cell. Conditions within the womb, such a maternal smoking, can have epigenetic effects. The investigators aim therefore to better understand how the environment experience by the fetus can affect development and programming of adult health and disease by epigenetic mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Women at 7-20 weeks of gestation (critical stage of fetal development).
* Women aged 16 years and older, deemed capable of making a rational decision.
* Absence of fetal anomaly at ultrasound scan (only normal fetuses are required).
* Women who are fluent English speakers. This is in order to ensure the woman understands that fetal tissues will be collected.

Exclusion Criteria:

* Women exhibiting considerable emotional distress.
* Fetal anomalies identified at ultrasound scan.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Human fetuses and their placentas collected without incentive from elective medical termination of normally progressing pregnancies. Data from the mothers is included in analyses.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
The provision of an extensive dataset on the human fetus during normal pregnancy and pregnancies where aspects of maternal lifestyle and environment will challenge the fetus, informing on future heath and function. | Whole project, up to 10 years
  The provision of an extensive dataset on the human fetus during normal pregnancy and pregnancies where aspects of maternal lifestyle and environment will challenge the fetus, informing on future heath and function.

SECONDARY OUTCOMES:
(1) The identification of key stages and regulators required for the normal development of the human fetus and its placenta. | Whole project, up to 10 years
  (1) The identification of key stages and regulators required for the normal development of the human fetus and its placenta.
(2) The quantification of maternal lifestyle factors, including body burdens of toxicant chemicals (e.g. from smoking, from air pollution, from food contact material) and determination of their relationship with adverse fetal and placental outcomes. | Whole project, up to 10 years
  (2) The quantification of maternal lifestyle factors, including body burdens of toxicant chemicals (e.g. from smoking, from air pollution, from food contact material) and determination of their relationship with adverse fetal and placental outcomes.
(3) Mechanistic insights into how fetal human development is controlled and how this control can be disturbed by maternal factors. | Whole project, up to 10 years
  (3) Mechanistic insights into how fetal human development is controlled and how this control can be disturbed by maternal factors.
(4) Establishment of the risks of adverse in-utero environment for future generations. This is epigenetic and focuses on ways in which fetal event, without any changes in genes themselves, can mis-programme the development of future generations. | Whole project, up to 10 years
  (4) Establishment of the risks of adverse in-utero environment for future generations. This is epigenetic and focuses on ways in which fetal event, without any changes in genes themselves, can mis-programme the development of future generations.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Fowler, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Result] Vazakidou P, Evangelista S, Li T, Lecante LL, Rosenberg K, Koekkoek J, Salumets A, Velthut-Meikas A, Damdimopoulou P, Mazaud-Guittot S, Fowler PA, Leonards PEG, van Duursen MBM. The profile of steroid hormones in human fetal and adult ovaries. Reprod Biol Endocrinol. 2024 May 22;22(1):60. doi: 10.1186/s12958-024-01233-7. PMID 38778396
- [Result] Bongaerts E, Lecante LL, Bove H, Roeffaers MBJ, Ameloot M, Fowler PA, Nawrot TS. Maternal exposure to ambient black carbon particles and their presence in maternal and fetal circulation and organs: an analysis of two independent population-based observational studies. Lancet Planet Health. 2022 Oct;6(10):e804-e811. doi: 10.1016/S2542-5196(22)00200-5. PMID 36208643
- [Result] Mamsen LS, Zafeiri A, Botkjaer JA, Hardlei JR, Ernst E, Oxvig C, Fowler PA, Andersen CY. Expression of the Insulin-like Growth Factor System in First- and Second-Trimester Human Embryonic and Fetal Gonads. J Clin Endocrinol Metab. 2020 Sep 1;105(9):e3157-68. doi: 10.1210/clinem/dgaa470. PMID 32726409
- [Result] Walker N, Filis P, O'Shaughnessy PJ, Bellingham M, Fowler PA. Nutrient transporter expression in both the placenta and fetal liver are affected by maternal smoking. Placenta. 2019 Mar;78:10-17. doi: 10.1016/j.placenta.2019.02.010. Epub 2019 Feb 25. PMID 30955705
- [Result] O'Shaughnessy PJ, Antignac JP, Le Bizec B, Morvan ML, Svechnikov K, Soder O, Savchuk I, Monteiro A, Soffientini U, Johnston ZC, Bellingham M, Hough D, Walker N, Filis P, Fowler PA. Alternative (backdoor) androgen production and masculinization in the human fetus. PLoS Biol. 2019 Feb 14;17(2):e3000002. doi: 10.1371/journal.pbio.3000002. eCollection 2019 Feb. PMID 30763313
- [Result] Johnston ZC, Bellingham M, Filis P, Soffientini U, Hough D, Bhattacharya S, Simard M, Hammond GL, King P, O'Shaughnessy PJ, Fowler PA. The human fetal adrenal produces cortisol but no detectable aldosterone throughout the second trimester. BMC Med. 2018 Feb 12;16(1):23. doi: 10.1186/s12916-018-1009-7. PMID 29429410

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT04613583/Prot_SAP_001.pdf
  • Informed Consent Form (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04613583/ICF_000.pdf